CLINICAL TRIAL: NCT02964728
Title: Botulinum Toxin in Burning Mouth Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Presidio Ospedaliero Garibaldi-Centro (Other)
Collaborators: Carlo Besta Neurological Institute (Other); University of Catania (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Domenico Antonio Restivo, MD, Presidio Ospedaliero Garibaldi-Centro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BMS-1
Record Dates: First submitted 2016-11-12; First posted 2016-11-16 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Burning Mouth Syndrome
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin type A (Experimental): Botulinum neurotoxin injections
  Interventions: Drug: Botulinum Neurotoxin Type A
- Placebo (Placebo Comparator): Normal saline solution injections
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Botulinum Neurotoxin Type A — topical injection
  Arms: Botulinum toxin type A
Other: Normal saline — topical injection
  Arms: Placebo

SUMMARY:
The effect of botulinum neurotoxin type A intradermal injection in will be evaluated in 4 patients with clinical diagnosis of burning mouth syndrome involving the anterior two-thirds of the tongue and the lower lip for at least 6 months, refractory to common pharmacological treatments. Pain severity will be measured by the visual analog scale (VAS) indicating average week pain before injection. Each patient will be injected with a total dose of 16 units (dilution: 2 ml saline) of incobotulinumA: 4 units into each side of the lower lip and 4 units into each antero-lateral side of the tongue. In order to determine if a placebo effect may be involved, we will inject 2 additional patients with saline solution using the same volumes and the same injection sites. Patients will be evaluated at 48 hours and then at 4, 8, 12, 16 and 20 weeks after the treatment. Patients treated with placebo will be treated after 4 weeks with incobotulinumA with the same dose reported above.

ELIGIBILITY:
Inclusion Criteria:

* burning mouth syndrome

Exclusion Criteria:

* any other mouth disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
0-100 mm Visual Analog Scale (VAS) improvement | 1 month

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lauria G, Majorana A, Borgna M, Lombardi R, Penza P, Padovani A, Sapelli P. Trigeminal small-fiber sensory neuropathy causes burning mouth syndrome. Pain. 2005 Jun;115(3):332-337. doi: 10.1016/j.pain.2005.03.028. PMID 15911160
- [Result] Ranoux D, Attal N, Morain F, Bouhassira D. Botulinum toxin type A induces direct analgesic effects in chronic neuropathic pain. Ann Neurol. 2008 Sep;64(3):274-83. doi: 10.1002/ana.21427. PMID 18546285
- [Result] Restivo DA, Tinazzi M, Patti F, Palmeri A, Maimone D. Botulinum toxin treatment of painful tonic spasms in multiple sclerosis. Neurology. 2003 Sep 9;61(5):719-20. doi: 10.1212/01.wnl.0000080081.74117.e4. No abstract available. PMID 12963779